CLINICAL TRIAL: NCT03399903
Title: Study of Pentasa® for Reducing Residual Systemic Immune Activation in Treated HIV Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AIDS Healthcare Foundation (Other)
Collaborators: HIV Immunotherapeutics Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HII-03
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: HIV-1-infection; Gut Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentasa (Experimental): 40 participants will be randomized to take 1 gram of Pentasa, twice daily for 8 weeks
  Interventions: Drug: Pentasa vs Align
- Align (Active Comparator): 40 participants will be randomized to take Align tablets, once daily for 8 weeks
  Interventions: Drug: Pentasa vs Align

INTERVENTIONS:
Drug: Pentasa vs Align — We will examine the safety and possible effectiveness of Pentasa® and Align in reducing markers of immune activation believed to be important reflectors of risk for cardiovascular disease and ongoing immune damage in people with chronic treated HIV-1 infection.

SUMMARY:
An open label study will be performed on 80 people with HIV infection who are maintained on effective treatment with antiretroviral drugs.

DETAILED DESCRIPTION:
The goal of this study is to test whether a bowel anti-inflammatory drug that is known to be safe and effective for inflammatory bowel disease would offer benefit in reducing the residual immune activation associated with treated HIV-1 infection. Specifically, the two immediate goals are to examine the safety of Pentasa® in reducing markers of immune activation believed to be important reflectors of risk for cardiovascular disease and ongoing immune damage in people with chronic treated HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18
* On ART for at least 1 year during which: viremia <50 RNA copies/ml for at least 3 measurements (allowing for 1 nonconsecutive blip of <100), and CD4 T cell count consistently >500 during that time
* CD4 T cell nadir >350
* Last CD4 and T cell test in past 6 months

Exclusion Criteria:

* Plans to modify antiretroviral therapy in the next 12 weeks for any reason
* History of inflammatory bowel disease or irritable bowel disease
* Chronic active hepatitis B or C
* History of autoimmune disease
* Hypersensitivity to any component of Pentasa
* Clostridium difficile infection
* Receiving rectally delivered medications
* Receiving anti-inflammatory medications (such as nonsteroidal anti- inflammatory drugs, steroids, or TNF inhibitors)
* Receiving immunosuppressive steroids
* Receiving any medications associated with bleeding risk
* Hemoglobin < 10.0 g/dL
* Platelet count less than 100,000/mm3
* White blood cell count < 2,000 cells/mm3 or > 15,000 cells/mm3
* Symptoms of sexually transmitted infection
* Antibiotics used in the last 90 days
* Renal insufficiency with creatinine clearance less than 50 ml/min
* Elevated transaminases greater than 2.5 times the upper limit of normal
* Evidence of decompensated cirrhosis, heart failure
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Inflammation markers | 14 weeks
  C-reactive protein

SECONDARY OUTCOMES:
Flow cytometry for cellular immune activation | 14 weeks
  Immune activation
Plasma markers of microbial translocation | 14 weeks
  Microbial translocation

CONTACTS AND LOCATIONS:
Overall Officials: Otto O Yang, MD, Study Director — AIDS Healthcare Foundation - HIV Immunotherapeutics Institute; Peter Anton, MD, Principal Investigator — AIDS Healthcare Foundation - HIV Immunotherapeutics Institute
Locations (1):
- AIDS Healthcare Foundation - Public Health Division, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No